CLINICAL TRIAL: NCT02713620
Title: Comparison of Immunogenicity of Four Doses and Four Double Doses vs. Standard Doses of Hepatitis B Vaccination in HIV-infected Adults: a Result From Randomized Controlled Trial at 3 Years After Vaccination
Brief Title: Hepatitis B Vaccination in HIV-infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Research ID: 2986
Record Dates: First submitted 2016-03-04; First posted 2016-03-21 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
Keywords: HBV vaccination, immunity
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy (Placebo Comparator): the "Healthy group" receiving three intramuscular injections of 20 μg of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, and 6
  Interventions: Biological: recombinant HBV vaccine (Hepavax-Gene® Berna, Korea)
- HIV-Group1 (Active Comparator): the "Standard doses group" receiving three intramuscular injections of 20 μg of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, and 6
  Interventions: Biological: recombinant HBV vaccine (Hepavax-Gene® Berna, Korea)
- HIV-Group 2 (Active Comparator): the "Four doses group" receiving four intramuscular doses of 20 μg of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, 2, and 6
  Interventions: Biological: recombinant HBV vaccine (Hepavax-Gene® Berna, Korea)
- HIV-Group 3 (Active Comparator): the "Four double doses group" receiving four intramuscular double doses (40 μg) of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, 2, and 6
  Interventions: Biological: recombinant HBV vaccine (Hepavax-Gene® Berna, Korea)

INTERVENTIONS:
Biological: recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) — Different HBV vaccine regimen in each group

SUMMARY:
This is a follow up study from the published article entitled "Comparison of immunogenicity and safety of four doses and four double doses vs. standard doses of hepatitis B vaccination in HIV-infected adults: a randomized, controlled trial" by Chaiklang K, Wipasa J, Chaiwarith R, Praparattanapan J, Supparatpinyo K. that was published in PLoS One. 2013 Nov 12;8(11):e80409. doi: 10.1371/journal.pone.0080409. eCollection 2013. ClinicalTrials.gov; NCT1289106. This study aimed to evaluate the efficacy of the HBV vaccination regimens using either four standard doses or four double doses compared with the current standard regimen of three doses in HIV-infected adults in northern Thailand. In addition, the investigators evaluated the efficacy of the HBV vaccination with the current standard regimen of three doses between healthy adults and HIV-infected patients.

DETAILED DESCRIPTION:
From February 4, 2011 to May 4, 2012, 132 HIV-infected adults with CD4+ cell counts >200 cells/mm3, undetectable plasma HIV-1 RNA, and negative for all HBV markers were randomly assigned to receive one of three recombinant vaccine (Hepavax-Gene® Berna, Korea) regimens: 20 μg IM at months 0, 1, and 6 (Standard doses group, n=44), 20 μg IM at months 0, 1, 2, 6 (four doses group, n=44), or 40 μg IM at months 0, 1, 2, and 6 (four double doses group, n=44). There was another group of healthy individuals received standard dose of 20 μg IM at months 0, 1, and 6 recruited during the same time and under the same protocol. In brief, at months 7 and 12, the percentages of responders (anti-HBs ≥10 mIU/mL) were 88.6% and 70.4% in the Standard doses group, 93.2% and 86.4% in the four doses group, (P=0.713 and 0.119), and 95.4% and 88.6% in the four double doses group, (P=0.434 and 0.062), respectively.

This current study aimed to evaluate the efficacy of the different HBV vaccination regimens at 36 months after vaccination. In addition to compare the group using four standard doses or four double doses with the current standard regimen of three doses in HIV-infected adults in northern Thailand, the investigators also compare the efficacy of the current standard regimen of 3 doses between HIV-infected and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Group 1.1 ≥18 years old, 1.2 were negative for hepatitis B surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc), had no history of previous vaccine 1.3 were negative for antibody to hepatitis C virus (anti-HCV) 1.4 received three intramuscular injections of 20 μg of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, and 6 during February 4, 2011 to May 4, 2012, the same time as the study under ClinicalTrials.gov; NCT1289106. were conducted.

   1.4 and were willing to sign an informed consent
2. HIV Group 1 2.1 HIV-1 infection 2.2 ≥18 years old, 2.3 had a CD4+ cell count >200 cells/mm3, 2.4 undetectable plasma HIV-1 RNA, 2.5 were negative for hepatitis B surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc), had no history of previous vaccine, 2.6 were negative for antibody to hepatitis C virus (anti-HCV), 2.7 had no active opportunistic infections (at the time of screening), 2.8 were participated in ClinicalTrials.gov; NCT1289106.and receiving three intramuscular injections of 20 μg of recombinant HBV vaccine (Hepavax-Gene® Berna, Korea) at months 0, 1, and 6 2.9 were willing to sign an informed consent
3. HIV-Group 2 3.1 HIV-1 infection 3.2 ≥18 years old, 3.3 had a CD4+ cell count >200 cells/mm3, 3.4 undetectable plasma HIV-1 RNA, 3.5 were negative for hepatitis B surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc), had no history of previous vaccine, 3.6 were negative for antibody to hepatitis C virus (anti-HCV), 3.7 had no active opportunistic infections (at the time of screening), 3.8 were participated in ClinicalTrials.gov; NCT1289106.and receiving four intramuscular doses of 20 μg of the same vaccine at months 0, 1, 2, and 6 3.9 were willing to sign an informed consent
4. HIV Group 3 4.1 HIV-1 infection 4.2 ≥18 years old, 4.3 had a CD4+ cell count >200 cells/mm3, 4.4 undetectable plasma HIV-1 RNA, 4.5 were negative for hepatitis B surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc), had no history of previous vaccine, 4.6 were negative for antibody to hepatitis C virus (anti-HCV), 4.7 had no active opportunistic infections (at the time of screening), 4.8 were participated in ClinicalTrials.gov; NCT1289106.and receiving four intramuscular double doses (40 μg) at months 0, 1, 2, and 6 4.9 were willing to sign an informed consent

Exclusion Criteria:

For HIV group 1, 2, and 3

1. active malignancy receiving chemotherapy or radiation,
2. other immunocompromised conditions besides HIV (e.g., solid organ transplant),
3. received immunosuppressive (e.g., corticosteroid ≥ 0•5 mg/kg/day) or immunomodulating treatment in the last six months before screening visit, 4. had renal insufficiency (creatinine clearance <30 mL/min), 5. decompensated cirrhosis (Child-Pugh class C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with protective immunity against HBV | 36 months after vaccination
  Comparison of proportion of participants who had protective immunity (anti-HBS titer >=10 mIU/ml) against HBV between "healthy" v.s. "HIV group 1", "HIV group 2" v.s. "HIV group 1", "HIV group 3 v.s. "HIV group 1"

SECONDARY OUTCOMES:
The geometric means of anti-HBs titers | 36 months after vaccination
  Comparison of the geometric means of anti-HBS titers between "healthy" v.s. "HIV group 1", "HIV group 2" v.s. "HIV group 1", "HIV group 3 v.s. "HIV group 1"
Proportion of participants with high level of immune response against HBV | 36 months after vaccination
  Comparison of proportion of participants who had anti-HBS titers >=100 mIU/ml between "healthy" v.s. "HIV group 1", "HIV group 2" v.s. "HIV group 1", "HIV group 3 v.s. "HIV group 1"

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Chiang Mai Unviersity
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaiwarith R, Praparattanapan J, Kotarathititum W, Wipasa J, Chaiklang K, Supparatpinyo K. Higher rate of long-term serologic response of four double doses vs. standard doses of hepatitis B vaccination in HIV-infected adults: 4-year follow-up of a randomised controlled trial. AIDS Res Ther. 2019 Nov 11;16(1):33. doi: 10.1186/s12981-019-0249-8. PMID 31711528